CLINICAL TRIAL: NCT02957994
Title: Analysis of Proximal Renal Tubular Function of "Real World" Chronic Hepatitis B (CHB) Patients Who Are Suppressed on TDF and Switched to TAF
Brief Title: TAF Switch Study in Hepatitis B Monoinfection
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Asian Pacific Liver Center at Coalition of Inclusive Medicine (Other)
Responsible Party: Principal Investigator, Ho Bae, Medical Director, Asian Pacific Liver Center at Coalition of Inclusive Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IN-US-320-4200
Record Dates: First submitted 2016-10-24; First posted 2016-11-08 (Estimated); Last update posted 2017-06-29 (Actual); Status verified 2017-06

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- TAF Arm (Experimental): Tenofovir alafenamide fumarate 25mg, 1 tablet once daily for 24 weeks
  Interventions: Drug: Tenofovir alafenamide fumarate

INTERVENTIONS:
Drug: Tenofovir alafenamide fumarate — Patients on TDF will be switched to TAF
  Other Names: TAF

SUMMARY:
To evaluate various markers of renal function and bone density after the switch to Tenofovir alafenamide fumarate (TAF) in chronic hepatitis B patients who are currently treated with Tenofovir disoproxil fumarate (TDF) .

DETAILED DESCRIPTION:
The investigators have previously reported the prevalence of abnormal renal tubular reabsorption of phosphate among CHB patients treated with more than 18 months of TDF to be 48%. Renal tubular dysfunction associated with TDF may be reversible when TDF is discontinued 4. Recently, TAF 25 mg daily was shown to have comparable efficacy to TDF 300 mg with respect to viral suppression in both HBeAg positive and HBeAg negative CHB patients (studies 110 and 108) at 48 weeks of therapy. As speculated, the systemic exposure to tenofovir was significantly less in patients exposed to TAF compared to those on TDF with strikingly less effects noted in a variety of renal and bone parameters for individuals receiving TAF. Notably, however, the question remains to what if any improvements may be seen in CHB patients switched from TDF to TAF.

The investigators propose a prospective open label study to evaluate various markers of renal function and bone density in 80 CHB patients who are currently treated with TDF who are switched to TAF.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic hepatitis B (who are either HBeAg reactive or non-reactive)
* Treated with TDF with unquantifiable Hepatitis B Virus (HBV) DNA by a sensitive Polymerase chain reaction (PCR) assay for a minimum of 6 months
* No prior nucleos(t)ide exposure prior to treatment with TDF
* Treatment with TDF for a minimum of 12 months

Exclusion Criteria:

* HIV Infection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2016-12-22 (Actual); Primary Completion 2017-06-21 (Actual); Study Completion 2017-11-01 (Estimated)

PRIMARY OUTCOMES:
measure renal function after switch to TAF | one year
  Kidney function will be measured by blood and urine to compare abnormal results before and after switching to TAF.
measure bone density after switch to TAF | one year
  Bone density will also be measured to compare T score and Z score before and after switching to TAF

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fong TL, Lee BT, Tien A, Chang M, Lim C, Ahn A, Bae HS. Improvement of bone mineral density and markers of proximal renal tubular function in chronic hepatitis B patients switched from tenofovir disoproxil fumarate to tenofovir alafenamide. J Viral Hepat. 2019 May;26(5):561-567. doi: 10.1111/jvh.13053. Epub 2019 Jan 16. PMID 30576085